CLINICAL TRIAL: NCT05601882
Title: A Phase 3b/4 Randomized, Open-label, Efficacy Assessor Blinded Study, Comparing the Safety and Assessor Blinded Efficacy of Upadacitinib to Dupilumab in Subjects With Moderate to Severe Atopic Dermatitis (Level-Up)
Brief Title: A Study to Evaluate Adverse Events and Change in Disease Activity Comparing Oral Upadacitinib to Subcutaneous Dupilumab in Adolescent and Adult Participants With Moderate to Severe Atopic Dermatitis
Acronym: Level Up
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M23-696; 2022-002482-15 (EudraCT Number)
Record Dates: First submitted 2022-10-31; First posted 2022-11-01 (Actual); Results first posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-01

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; AD; Level-Up; Upadacitinib; Dupilumab; RINVOQ
MeSH Terms: conditions — Dermatitis, Atopic | interventions — dupilumab; upadacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Dupilumab (Period 1) (Experimental): Adult participants received a loading dose of 600 mg dupilumab by subcutaneous (SC) injection at the Baseline visit followed by 300 mg dupilumab SC every other week (EOW) until Week 16.
  Adolescents (12 to 17 years of age and weighing at least 40 kg) received treatment according to their body weight. Participants weighing 40 to < 60 kg received a loading dose of 400 mg dupilumab SC at the Baseline visit followed by 200 mg SC EOW until Week 16. Those weighing 60 kg or more received a loading dose of 600 mg dupilumab SC at the Baseline visit followed by 300 mg dupilumab SC EOW until Week 16.
  Interventions: Drug: Dupilumab
- Upadacitinib (Period 1) (Experimental): Participants received 15 mg upadacitinib orally once a day (QD) up to Week 16. Starting at Week 4, participants had their dose increased to 30 mg QD if they had a < 50% reduction from Baseline in Eczema Area and Severity Index (EASI 50) response or a < 4-point improvement from Baseline in Worst Pruritus Numerical Rating Scale (WP-NRS; weekly average). Starting at Week 8, participants had their dose increased to 30 mg QD if they had a < EASI 75 response.
  Interventions: Drug: Upadacitinib
- Dupilumab -> Upadacitinib (Period 2) (Experimental): At Week 16, participants receiving dupilumab as per its label in Period 1 were reassigned based on their Eczema Area and Severity Index (EASI) response. Those with < EASI 75 were offered the option to receive oral doses of upadacitinib 15 mg QD in Period 2 up to Week 32. Those with ≥ EASI 75 completed the end of study procedures. Starting at Week 20, participants with < EASI 75 or a < 4-point improvement from Baseline in Worst Pruritus Numerical Rating Scale (WP-NRS; weekly average) had their dose increased to 30 mg QD up to Week 32.
  Interventions: Drug: Upadacitinib
- Upadacitinib -> Upadacitinib 30 mg (Period 2) (Experimental): At Week 16, participants receiving upadacitinib in Period 1 were reassigned based on their Eczema Area and Severity Index (EASI) response. Those with < EASI 75 were allocated or continued to receive upadacitinib 30 mg QD in Period 2. Those with ≥ EASI 75 completed the end of study procedures.
  Interventions: Drug: Upadacitinib

INTERVENTIONS:
Drug: Dupilumab — Dupilumab is administered as a subcutaneous (SC) injection.
  Other Names: Dupixent®
  Arms: Dupilumab (Period 1)
Drug: Upadacitinib — Extended-release tablet
  Other Names: ABT-494; RINVOQ
  Arms: Dupilumab -> Upadacitinib (Period 2); Upadacitinib (Period 1); Upadacitinib -> Upadacitinib 30 mg (Period 2)

SUMMARY:
Atopic dermatitis (AD) is a skin condition that may cause a rash and itching due to inflammation of the skin. Therapies spread over the skin may not be enough to control the AD in trial participants who require systemic anti-inflammatory treatment. This study compares upadacitinib to dupilumab in adolescent and adult participants with moderate to severe AD who have inadequate response to systemic therapies. Adverse events and change in the disease activity will be assessed.

Upadacitinib and dupilumab are approved drugs for the treatment of moderate to severe atopic dermatitis (AD). The study is comprised of a 35-day Screening Period, a 16-week treatment Period 1 and a 16-week treatment Period 2. Participants are randomly assigned to 1 of 2 groups called treatment arms to receive upadacitinib Dose A or dupilumab in Period 1. There is a 30-day or 12-week follow-up visit for those on upadacitinib or dupilumab respectively, who will not enter Period 2. In Period 2, participants will receive upadacitinib Dose A or Dose B for 16 weeks, followed by a 30-day follow-up visit. Approximately 880 adolescent and adult participants ages 12 to 64 with moderate to severe AD who are candidates for systemic therapy will be enrolled at up to 330 sites worldwide.

There may be higher treatment burden for participants in this trial compared to their standard of care . Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Chronic atopic dermatitis (AD) with onset of symptoms at least 3 years prior to baseline and participant meets Hanifin and Rajka criteria.
* Eczema area and severity index (EASI) score ≥ 16;validated Investigator´s Global Assessment for AD (vIGA-AD) score ≥ 3 and ≥ 10% Body Surface Area Involvement of Atopic Dermatitis (BSA of AD) involvement at the Baseline Visit.
* Baseline weekly average of daily Worst Pruritus Numerical Rating Scale (WP-NRS) ≥ 4.
* Documented history of inadequate response to previous systemic treatment defined as documented history of previous inadequate response to at least one prior systemic treatment for AD OR for whom other systemic treatments are otherwise medically inadvisable.

Exclusion Criteria:

* History of clinically significant (per investigator's judgment) drug or alcohol abuse within the last 6 months.
* History of an organ transplant which requires continued immunosuppression.

Ages: 12 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 920 (Actual)
Dates: Start 2022-11-28 (Actual); Primary Completion 2024-03-19 (Actual); Study Completion 2024-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (257):
- United States (58):
  - Medical Dermatology Specialists /ID# 250212, Phoenix, Arizona
  - Alliance Dermatology and Mohs Center /ID# 249671, Phoenix, Arizona
  - Clinical Trials Institute - Northwest Arkansas /ID# 249838, Fayetteville, Arkansas
  - Arkansas Research Trials /ID# 250722, North Little Rock, Arkansas
  - Joseph Raoof Md,Inc /Id# 250211, Encino, California
  - First OC Dermatology /ID# 250686, Fountain Valley, California
  - Antelope Valley Clinical Trials /ID# 249946, Lancaster, California
  - Dermatology Research Associates /ID# 249829, Los Angeles, California
  - University of California Davis Health /ID# 250044, Sacramento, California
  - Clinical Trials Research Institute /ID# 250213, Thousand Oaks, California
  - Western States Clinical Res /ID# 250274, Wheat Ridge, Colorado
  - UConn Health /ID# 253807, Farmington, Connecticut
  - Yale Center for Clinical Investigation /ID# 254791, New Haven, Connecticut
  - Clearlyderm Dermatology /ID# 250457, Boca Raton, Florida
  - Skin Care Research Boca Raton /ID# 250458, Boca Raton, Florida
  - Olympian Clinical Research /ID# 250453, Clearwater, Florida
  - Skin Care Research - Hollywood /ID# 250459, Hollywood, Florida
  - Solutions Through Adv Rch /ID# 250455, Jacksonville, Florida
  - GSI Clinical Research, LLC /ID# 250768, Margate, Florida
  - D&H National Research Centers /ID# 250734, Miami, Florida
  - Florida International Rsrch cr /ID# 249667, Miami, Florida
  - Wellness Clinical Research - Miami Lakes /ID# 250236, Miami Lakes, Florida
  - Tory P Sullivan, MD PA /ID# 251136, North Miami Beach, Florida
  - Precision Clinical Research /ID# 250990, Sunrise, Florida
  - Advanced Clinical Research Institute /ID# 250460, Tampa, Florida
  - Metabolic Research Inst /ID# 250046, West Palm Beach, Florida
  - Treasure Valley Medical Research /ID# 250727, Boise, Idaho
  - Dawes Fretzin, LLC /ID# 250276, Indianapolis, Indiana
  - Randall Dermatology of West Lafayette /ID# 250234, West Lafayette, Indiana
  - Beth Israel Deaconess Medical Center /ID# 251212, Boston, Massachusetts
  - Beacon Clinical Research, LLC /ID# 251412, Quincy, Massachusetts
  - Clarkston Dermatology /ID# 250225, Clarkston, Michigan
  - Henry Ford Medical Center - New Center One /ID# 250228, Detroit, Michigan
  - Cleaver Dermatology /ID# 250725, Kirksville, Missouri
  - MediSearch Clinical Trials /ID# 250272, Saint Joseph, Missouri
  - Duplicate_Allergy, Asthma & Immunology Associates, PC /ID# 250616, Lincoln, Nebraska
  - Physician Research Collaboration, LLC /ID# 251099, Lincoln, Nebraska
  - Montefiore Medical Center - Moses Campus /ID# 251214, The Bronx, New York
  - Derm of Greater Columbus /ID# 250049, Bexley, Ohio
  - Univ Hosp Cleveland /ID# 250699, Cleveland, Ohio
  - Wright State Physicians - Fairborn /ID# 254167, Fairborn, Ohio
  - Vital Prospects Clinical Research Institute, PC /ID# 249840, Tulsa, Oklahoma
  - Oregon Dermatology and Research Center /ID# 250726, Portland, Oregon
  - Oregon Medical Research Center /ID# 249666, Portland, Oregon
  - Oregon Medical Research Center /ID# 250712, Portland, Oregon
  - University of Pittsburgh MC /ID# 251208, Pittsburgh, Pennsylvania
  - Duplicate_Medical University of South Carolina /ID# 251218, Charleston, South Carolina
  - Health Concepts /ID# 250988, Rapid City, South Dakota
  - International Clinical Research - Tennessee LLC /ID# 250724, Murfreesboro, Tennessee
  - Arlington Research Center, Inc /ID# 250468, Arlington, Texas
  - Orion Clinical Research /ID# 250473, Austin, Texas
  - Bellaire Dermatology Associates /ID# 250739, Bellaire, Texas
  - Modern Research Associates, PLLC /ID# 250688, Dallas, Texas
  - Center for Clinical Studies - Houston - Northwest Freeway /ID# 250039, Houston, Texas
  - Texas Dermatology and Laser Specialists /ID# 250367, San Antonio, Texas
  - University of Utah /ID# 250042, Murray, Utah
  - University of Virginia - Dermatology /ID# 254166, Charlottesville, Virginia
  - Virginia Clinical Research, Inc. /ID# 249908, Norfolk, Virginia
- Australia (5):
  - Premier Specialist /ID# 250572, Kogarah, New South Wales
  - Veracity Clinical Research /ID# 249943, Woolloongabba, Queensland
  - Skin Health Institute Inc /ID# 249938, Carlton, Victoria
  - Sinclair Dermatology - Melbourne /ID# 249937, East Melbourne, Victoria
  - Fremantle Dermatology /ID# 249941, Fremantle, Western Australia
- Belgium (4):
  - Cliniques Universitaires UCL Saint-Luc /ID# 251403, Woluwe-Saint-Lambert, Brussels Capital
  - Grand Hopital de Charleroi /ID# 251401, Charleroi, Hainaut
  - Universitair Ziekenhuis Leuven /ID# 251399, Leuven, Vlaams-Brabant
  - CHU de Liege /ID# 251400, Liège
- Bulgaria (9):
  - UMHAT Dr Georgi Stranski EAD /ID# 251268, Pleven, Smolyan
  - Diagnostic Consultative Center Aleksandrovska /ID# 251137, Sofiya, Sofia
  - DCC Pulmed AD /ID# 251271, Plovdiv
  - Ambulatory for Specialized Medical Care for skin and venereal diseases /ID# 251272, Sofia
  - Diagnostic consultative center Focus-5 /ID# 251269, Sofia
  - Medical Center Euroderma /ID# 251267, Sofia
  - Medical center EuroHealth /ID# 251270, Sofia
  - Military Medical Academy Multiprofile Hospital /ID# 251187, Sofia
  - MC Zara-Med EOOD /ID# 251135, Stara Zagora
- Canada (16):
  - Dermatology Research Institute - Blackfoot Trail /ID# 251642, Calgary, Alberta
  - Beacon Dermatology Inc /ID# 250336, Calgary, Alberta
  - Alberta DermaSurgery Centre /ID# 250217, Edmonton, Alberta
  - Dr. Chih-ho Hong Medical Inc. /ID# 251643, Surrey, British Columbia
  - Enverus Medical Research /ID# 251645, Surrey, British Columbia
  - Wiseman Dermatology Research /ID# 250219, Winnipeg, Manitoba
  - Brunswick Dermatology Center /ID# 250220, Fredericton, New Brunswick
  - LEADER Research /ID# 251647, Hamilton, Ontario
  - DermEffects /ID# 250223, London, Ontario
  - Lynde Institute for Dermatology /ID# 251854, Markham, Ontario
  - DermEdge Research Inc. /ID# 250216, Mississauga, Ontario
  - SKiN Centre for Dermatology /ID# 251853, Peterborough, Ontario
  - Toronto Dermatology Centre /ID# 252098, Toronto, Ontario
  - Research Toronto /ID# 250222, Toronto, Ontario
  - Private Practice - Dr. Kim Papp Clinical Research /ID# 251644, Waterloo, Ontario
  - Centre de Recherche dermatologique du Quebec Metropolitain /ID# 250427, Québec, Quebec
- China (14):
  - The First Affiliated Hospital Of Fujian Medical University /ID# 249674, Fuzhou, Fujian
  - Dermatology Hospital of Southern Medical University /ID# 250121, Guangzhou, Guangdong
  - Guangzhou First People's Hospital /ID# 249695, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Guangzhou Medical University /ID# 249694, Guangzhou, Guangdong
  - The University of Hong Kong- Shenzhen Hospital /ID# 249436, Shenzhen, Guangdong
  - The Second Xiangya Hospital of Central South University /ID# 249657, Changsha, Guizhou
  - Union Hospital Tongji Medical College Huazhong University of Science and Technol /ID# 251485, Wuhan, Hubei
  - The First Hospital of China Medical University /ID# 249638, Shenyang, Liaoning
  - Huashan Hospital, Fudan University /ID# 250025, Shanghai, Shanghai Municipality
  - Shanghai Skin Disease Hospital /ID# 249392, Shanghai, Shanghai Municipality
  - Tianjin Medical University General Hospital /ID# 250246, Tianjin, Tianjin Municipality
  - Hangzhou First People's Hospital /ID# 249437, Hangzhou, Zhejiang
  - The second affiliated hospital of Zhejiang University school of medicine /ID# 249655, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital /ID# 249653, Hangzhou, Zhejiang
- Croatia (7):
  - Poliklinika Solmed /ID# 252138, Grad Zagreb, City of Zagreb
  - DermaPlus - Poliklinika za dermatologiju i venerologiju /ID# 249591, Zagreb, City of Zagreb
  - Djecja bolnica Srebrnjak /ID# 249594, Zagreb, City of Zagreb
  - Klinicki bolnicki centar Zagreb /ID# 249596, Zagreb, City of Zagreb
  - Klinika za dječje bolesti Zagreb /ID# 249590, Zagreb, City of Zagreb
  - Klinicki bolnicki centar Rijeka /ID# 249593, Rijeka, Primorje-Gorski Kotar County
  - Klinicki Bolnicki Centar (KBC) Split /ID# 249879, Split, Split-Dalmatia County
- Denmark (4):
  - Bispebjerg and Frederiksberg Hospital /ID# 248902, Copenhagen NV, Capital Region
  - Herlev and Gentofte Hospital /ID# 248900, Hellerup, Capital Region
  - Aarhus Universitetshospital - Skejby /ID# 248899, Aarhus, Central Jutland
  - Roskilde Sygehus /ID# 248901, Roskilde, Region Sjælland
- France (6):
  - Hopital Saint Joseph /ID# 251053, Marseille, Bouches-du-Rhone
  - CHU de Nantes, Hotel Dieu -HME /ID# 251347, Nantes, Pays de la Loire Region
  - HCL - Hopital Lyon Sud /ID# 251343, Pierre-Bénite, Rhone
  - Hôpital Saint-Louis /ID# 251052, Paris
  - Hôpital Charles-Nicolle /ID# 251055, Rouen
  - CHU Toulouse - Hopital Larrey /ID# 251344, Toulouse
- Germany (19):
  - Universitaetsklinikum Freiburg /ID# 249555, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitaetsklinik Heidelberg /ID# 251458, Heidelberg, Baden-Wurttemberg
  - Universitaetsklinikum Tuebingen /ID# 249552, Tübingen, Baden-Wurttemberg
  - Dermatologische Gemeinschaftspraxis Mahlow /ID# 250306, Blankenfelde-Mahlow, Brandenburg
  - Klinikum Darmstadt /ID# 251391, Darmstadt, Hesse
  - Universitaetsklinikum Frankfurt /ID# 249544, Frankfurt am Main, Hesse
  - Studienzentrum an der Hase GbR Dr. Weyergraf/Dr. Frick/Thomas Heiber /ID# 251392, Bramsche, Lower Saxony
  - Universitaetsklinikum Bonn /ID# 250307, Bonn, North Rhine-Westphalia
  - Universitaetsklinikum Muenster /ID# 249404, Münster, North Rhine-Westphalia
  - Universitaetsmedizin Mainz /ID# 249549, Mainz, Rhineland-Palatinate
  - Fachklinik Bad Bentheim /ID# 249545, Bad Bentheim, Saarland
  - Universitaetsklinikum Leipzig /ID# 249562, Leipzig, Saxony
  - Universitaetsklinikum Schleswig-Holstein Campus Luebeck /ID# 249560, Lübeck, Schleswig-Holstein
  - Hautarztpraxis Dr. Niesmann und Dr. Othlinghaus /ID# 251566, Bochum
  - Universitaetsklinikum Carl Gustav Carus an der TU Dresden /ID# 251844, Dresden
  - Derma Study Center Friedrichshafen GmbH /ID# 251460, Friedrichshafen
  - Universitaetsklinikum Hamburg-Eppendorf /ID# 249547, Hamburg
  - Dermatologikum Hamburg /ID# 251390, Hamburg
  - Klinikum rechts der Isar /ID# 249548, Munich
- Greece (3):
  - 401 GSNA - 401 Army General Hospital /ID# 251843, Athens, Attica
  - General Hospital Andreas Syggros /ID# 251842, Athens, Attica
  - Papageorgiou General Hospital /ID# 251840, Thessaloniki, Evrytania
- Hungary (11):
  - Bacs-Kiskun Varmegyei Oktatokorhaz /ID# 249850, Kecskemét, Bács-Kiskun county
  - Debreceni Egyetem-Klinikai Kozpont /ID# 249849, Debrecen, Hajdú-Bihar
  - Gyongyosi Bugat Pal Korhaz /ID# 251367, Gyöngyös, Heves County
  - Pecsi Tudomanyegyetem Klinikai Kozpont /ID# 250419, Pecs, Nógrád megye
  - Somogy Varmegyei Kaposi Mor Oktato Korhaz /ID# 249848, Kaposvár, Somogy County
  - Clinexpert Kft /ID# 249822, Budapest
  - Semmelweis Egyetem /ID# 251368, Budapest
  - UNO Medical Trials /ID# 249820, Budapest
  - DERMA-B Egeszsegugyi es Szolgaltato - Debrecen - Gyepusor Utca /ID# 249819, Debrecen
  - Szegedi Tudományegyetem /ID# 249818, Szeged
  - Allergo-Derm Bakos Kft. /ID# 249821, Szolnok
- Israel (2):
  - Hadassah Medical Center-Hebrew University /ID# 251576, Jerusalem, Jerusalem
  - Rabin Medical Center /ID# 251578, Haifa
- Italy (12):
  - CAST - Center for Advanced Studies and Technology /ID# 251495, Chieti, L Aquila
  - Presidio Ospedaliero San Salvatore /ID# 250127, L’Aquila, L Aquila
  - IRCCS Istituto Clinico Humanitas /ID# 251493, Rozzano, Milano
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata /ID# 250125, Rome, Roma
  - IRCCS Istituti Fisioterapici Ospitalieri-Istituto Dermatologico San Gallicano /ID# 250558, Rome, Roma
  - Policlinico Agostino Gemelli /ID# 251494, Rome, Roma
  - ASST degli Spedali Civili di Brescia /ID# 250129, Brescia
  - Ospedale Piero Palagi /ID# 250206, Florence
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico /ID# 250123, Milan
  - Azienda Ospedaliero-Universitaria di Modena /ID# 250128, Modena
  - Azienda Ospedaliera di Perugia - Ospedale S. Maria della Misericordia /ID# 251572, Perugia
  - Azienda Ospedaliero Universitaria Pisana /ID# 250124, Pisa
- Japan (7):
  - Medical Corporation Kojinkai Sapporo Skin Clinic /ID# 252549, Sapporo, Hokkaido
  - Medical corporation Kojunkai Kosugi Dermatology Clinic /ID# 252554, Kawasaki-shi, Kanagawa
  - National Hospital Organization Sagamihara National Hospital /ID# 254518, Sagamihara-shi, Kanagawa
  - Queen's Square Medical Center, Dermatology and Allergology /ID# 252551, Yokohama, Kanagawa
  - Osaka Habikino Medical Center /ID# 252550, Habikino-shi, Osaka
  - Dermatology and Ophthalmology Kume Clinic /ID# 254570, Sakai-shi, Osaka
  - Naoko Dermatology Clinic /ID# 254571, Setagaya-ku, Tokyo
- Mexico (5):
  - Centro de Dermatologia de Monterrey /ID# 249126, Monterrey, Estado de Baja California
  - Eukarya PharmaSite, SC /ID# 249702, Monterrey, Nuevo León
  - Cryptex Investigacion Clinica S.A de C.V /ID# 249994, Mexico City
  - Clinical Research Institute SC /ID# 249647, Tlalnepantla
  - Arké Estudios Clinicos Veracruz /ID# 250147, Veracruz
- Netherlands (2):
  - Bravis Ziekenhuis /ID# 251395, Bergen op Zoom, North Brabant
  - Amsterdam UMC, locatie AMC /ID# 251397, Amsterdam, North Holland
- Poland (13):
  - Solumed Centrum Medyczne /ID# 249641, Poznan, Greater Poland Voivodeship
  - MICS Centrum Medyczne Torun /ID# 251433, Torun, Kuyavian-Pomeranian Voivodeship
  - Lidia Rajzer - Specjalistyczny Gabinet Dermatologiczno-Kosmetyczny /ID# 252082, Krakow, Lesser Poland Voivodeship
  - Centrum Nowoczesnych Terapii Dobry Lekarz Sp. z o.o. /ID# 251437, Krakow, Lesser Poland Voivodeship
  - Klinika Ambroziak Sp. z o.o. /ID# 249406, Warsaw, Masovian Voivodeship
  - Royalderm Agnieszka Nawrocka /ID# 251432, Warsaw, Masovian Voivodeship
  - Bodyclinic Sp. z o.o. sp.k. /ID# 249599, Warsaw, Masovian Voivodeship
  - Zespol Naukowo-Leczniczy Iwolang Dermatologiczne Centrum Uzdrowiskowe Sp. z o.o /ID# 249598, Iwonicz-Zdrój, Podkarpackie Voivodeship
  - INTER CLINIC Piotr Adrian Klimiuk /ID# 251430, Bialystok, Podlaskie Voivodeship
  - Centrum Badan Klinicznych PI-House sp. z o.o. /ID# 251431, Gdansk, Pomeranian Voivodeship
  - Centrum Kliniczno-Badawcze J.Brzezicki, B. Gornikiewicz-Brzezicka Lekarze Spolka /ID# 251438, Elblag, Warmian-Masurian Voivodeship
  - Centrum Medyczne ALL-MED Badania Kliniczne /ID# 249630, Krakow
  - Dermed Centrum Medyczne Sp. z o.o /ID# 251429, Lodz, Łódź Voivodeship
- Portugal (9):
  - Centro Hospitalar Do Alto Ave - Hospital Senhora Da Oliveira /ID# 249196, Guimarães, Braga District
  - Hospital CUF Descobertas /ID# 249193, Lisboa, Madeira
  - Centro Hospitalar Universitario do Porto, EPE - Hospital Santo Antonio /ID# 249191, Porto, Madeira
  - Hospital Garcia de Orta /ID# 251455, Almada, Setúbal District
  - 2CA-Braga, Hospital de Braga /ID# 250480, Braga
  - Unidade Local de Saude da Regiao de Leiria, EPE /ID# 249194, Leiria
  - Centro Hospitalar de Lisboa Central /ID# 249195, Lisbon
  - Unidade Local de Saúde de Matosinhos, EPE /ID# 249197, Matosinhos Municipality
  - Centro Hospitalar Universitario de Sao Joao, EPE /ID# 249192, Porto
- Puerto Rico (4):
  - Dr. Samuel Sanchez PSC /ID# 250389, Caguas
  - Alma M. Cruz Santana, MD-Private practice /ID# 250393, Carolina
  - Clinical Research Puerto Rico /ID# 250394, San Juan
  - GCM Medical Group PSC /ID# 250391, San Juan
- Romania (2):
  - Bio Terra Med SRL /ID# 249624, Bucharest, București
  - Private Practice - Dr. Orasan Remus /ID# 249625, Cluj-Napoca, Cluj
- Slovakia (3):
  - Derma therapy spol /ID# 249783, Bratislava, Bratislava Region
  - Poliklinika Bezrucova (Cliniq s.r.o.) /ID# 249746, Bratislava
  - BeneDerma s.r.o. /ID# 251791, Bratislava
- South Africa (5):
  - University of Pretoria /ID# 250208, Pretoria, Gauteng
  - About Allergy /ID# 249697, Pretoria, Gauteng
  - Highway Medical Centre /ID# 250103, Durban, KwaZulu-Natal
  - Allergy & Immunology (AIU) /ID# 249619, Cape Town, Western Cape
  - Spoke Research Inc /ID# 250091, CAPE TOWN Milnerton, Western Cape
- South Korea (8):
  - Pusan National University Hospital /ID# 249852, Busan, Busan Gwang Yeogsi
  - Kyungpook National University Hospital /ID# 249855, Junggu, Daegu Gwang Yeogsi
  - Korea University Ansan Hospital /ID# 249814, Ansan-si, Gyeonggido
  - Soon Chun Hyang University Hospital Bucheon /ID# 249812, Bucheon-si, Gyeonggido
  - Chungang University Hospital /ID# 251490, Dongjak-gu, Gyeonggido
  - Ajou University Hospital /ID# 251491, Suwon, Gyeonggido
  - Seoul National University Hospital /ID# 251492, Seoul, Seoul Teugbyeolsi
  - Konkuk University Medical Center /ID# 249811, Seoul, Seoul Teugbyeolsi
- Spain (8):
  - Hospital Universitario Germans Trias i Pujol /ID# 251523, Badalona, Barcelona
  - Hospital Sant Joan de Deu /ID# 249602, Esplugues de Llobregat, Barcelona
  - Hospital Universitario Basurto /ID# 249784, Bilbao, Vizcaya
  - Hospital General Universitario de Alicante Doctor Balmis /ID# 251517, Alicante
  - Hospital Universitario Virgen de las Nieves /ID# 249785, Granada
  - Hospital Universitario La Paz /ID# 251518, Madrid
  - Hospital Universitario Virgen Macarena /ID# 249603, Seville
  - Hospital Universitario y Politecnico La Fe /ID# 251524, Valencia
- Sweden (4):
  - Skane University hospital /ID# 250332, Malmo, Skåne County
  - Karolinska University Hospital Solna /ID# 250328, Solna, Stockholm County
  - Norrlands University hospital /ID# 250329, Umeå, Västerbotten County
  - Malarsjukhuset /ID# 251908, Eskilstuna
- Switzerland (2):
  - Kantonsspital St. Gallen /ID# 250606, Sankt Gallen, Canton of St. Gallen
  - Inselspital, Universitaetsspital Bern /ID# 250577, Bern
- Taiwan (9):
  - Kaohsiung Chang Gung Memorial Hospital /ID# 249260, Kaohsiung City, Kaohsiung
  - Taichung Veterans General Hospital /ID# 249261, Taichung, Keelung
  - National Taiwan University Hospital /ID# 249258, Taipei City, Taipei
  - National Taiwan University Hospital - Hsinchu branch /ID# 249265, Hsinchu
  - Taipei Medical University Shuang Ho Hospital /ID# 249256, New Taipei City
  - Mackay Memorial Hospital /ID# 249259, Taipei
  - Taipei Veterans General Hosp /ID# 249263, Taipei
  - Taipei Municipal Wan Fang Hospital /ID# 251500, Taipei
  - Linkou Chang Gung Memorial Hospital /ID# 249257, Taoyuan
- Turkey (Türkiye) (6):
  - Gaziantep Universitesi /ID# 249868, Gaziantep, Adana
  - Ankara City Hospital /ID# 249870, Ankara
  - Akdeniz Universitesi Tip Fakul /ID# 249866, Antalya
  - Uludag University Medical Faculty /ID# 249864, Bursa
  - Erciyes University Medical Faculty /ID# 249863, Kayseri
  - Ondokuz Mayis Universitesi /ID# 249865, Samsun

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Bunick CG, Magnolo N, Moore A, Abe M, Gao X, Lynde C, Ibrahim N, Levy G, Calimlim BM, Wu X, Armendariz Y, Grada A, Eyerich K. Switching from Dupilumab to Upadacitinib in Adults and Adolescents with Moderate-to-Severe Atopic Dermatitis After Inadequate Response to Dupilumab: Efficacy and Safety Results from Period 2 of Phase 3b/4 Study (LEVEL UP). Am J Clin Dermatol. 2026 Jan 14. doi: 10.1007/s40257-025-01003-0. Online ahead of print. PMID 41533220
- See also: Related info — https://www.rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized at 214 sites located in 28 countries (Australia, Belgium, Bulgaria, Canada, China, Croatia, Denmark, France, Germany, Greece, Hungary, Israel, Italy, Japan, Korea, Mexico, Netherlands, Poland, Portugal, Romania, Slovakia, South Africa, Spain, Sweden, Switzerland, Taiwan, Turkey, and the United States/Puerto Rico).
Pre-assignment Details: Participants who met eligibility criteria were randomized in a 1:1 ratio to receive either upadacitinib 15 mg QD or dupilumab as per its label in Period 1. At Week 16, participants from both Period 1 arms with a < EASI 75 response entered Period 2; those from the dupilumab arm were offered the option to receive upadacitinib 15 mg QD while those from the upadacitinib arm either continued (if already receiving 30 mg) or escalated to upadacitinib 30 mg QD (if receiving 15 mg QD) until Week 32.
Period: Period 1 (Baseline - Week 16)
Arm/Group | Dupilumab (Period 1) | Upadacitinib (Period 1) | Dupilumab -> Upadacitinib (Period 2) | Upadacitinib -> Upadacitinib 30 mg (Period 2)
Started | 462 | 458 | 0 | 0
Completed | 423 | 418 | 0 | 0
Not Completed | 39 | 40 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 21 | 24 | 0 | 0
Not completed — Other, not specified | 16 | 16 | 0 | 0
Period: Period 2 (Week 16 - Week 32)
Arm/Group | Dupilumab (Period 1) | Upadacitinib (Period 1) | Dupilumab -> Upadacitinib (Period 2) | Upadacitinib -> Upadacitinib 30 mg (Period 2)
Started | 0 | 0 | 208 | 147
Completed | 0 | 0 | 198 | 131
Not Completed | 0 | 0 | 10 | 16
Not completed — Lost to Follow-up | 0 | 0 | 3 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 3 | 4
Not completed — Other, not specified | 0 | 0 | 4 | 11

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population of Period 1 (ITT_1 Population): all participants who were randomized at Baseline, analyzed per the treatment group to which they were randomized
Groups:
- Total: Total of all reporting groups
Arm/Group | Dupilumab (Period 1) | Upadacitinib (Period 1) | Total
Number analyzed (Participants) | 462 | 458 | 920
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.9 (12.79) | 31.0 (12.71) | 31.0 (12.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 217 | 195 | 412
  Male | 245 | 263 | 508
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 41 | 44 | 85
  Not Hispanic or Latino | 421 | 414 | 835
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 137 | 122 | 259
  Native Hawaiian or Other Pacific Islander | 1 | 3 | 4
  Black or African American | 19 | 20 | 39
  White | 296 | 303 | 599
  More than one race | 5 | 6 | 11
  Unknown or Not Reported | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving a ≥ 90% Reduction From Baseline in Eczema Area and Severity Index Score (EASI 90) and Worst Pruritus Numerical Rating Scale of 0 or 1 (WP-NRS 0/1) at Week 16
Description: The EASI is a composite index with scores ranging from 0 to 72. Four AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) assessed for severity on a scale of "0" (absent) through "3" (severe). In addition, the area of AD involvement is assessed as a percentage by body area of head, trunk (including the genital area), upper extremities, and lower extremities (including the buttocks), and converted to a score of 0 to 6. In each body region, the area is expressed as 0, 1 (1% to 9%), 2 (10% to 29%), 3 (30% to 49%), 4 (50% to 69%), 5 (70% to 89%), or 6 (90% to 100%).
  The Worst Pruritus NRS is an assessment tool that participants used to report the intensity of their pruritus during a 24-hour recall period using an electronic hand-held device. Participants rated itch (pruritus) intensity at its worst during the past 24 hours on an 11-point scale from 0 (no itch) to 10 (worst imaginable itch).
Time Frame: Baseline and Week 16
Population: Intent-to-Treat (ITT) Population of Period 1 (ITT_1 Population): all participants who were randomized at Baseline; non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 or any other missing data that can be reasonably assumed to be Missing at Random (NRI-MI) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dupilumab (Period 1) | Upadacitinib (Period 1)
Number analyzed (Participants) | 462 | 458
percentage of participants | 8.9 [6.3 to 11.5] | 19.9 [16.2 to 23.5]
Statistical Analysis 1: Comparison: Dupilumab (Period 1) vs Upadacitinib (Period 1); Upadacitinib (Period 1) vs Dupilumab (Period 1); Test type: Superiority — Analyzed using Cochran-Mantel-Haenszel (CMH) test stratified by Validated Investigator's Global Assessment for Atopic Dermatitis categories [(vIGA-AD (moderate [3] versus severe [4])] and age (12 to < 18; 18 to < 40; ≥40 to < 64 years); p < 0.0001, Cochran-Mantel-Haenszel; Adjusted Response Rate Difference = 11.0, 95% CI 2-sided [6.6 to 15.5] — Response rate difference = Upadacitinib (Period 1) - Dupilumab (Period 1)

2. Secondary Outcome: Percentage of Participants Achieving a ≥ 90% Reduction From Baseline in Eczema Area and Severity Index Score (EASI 90) at Week 16
Description: The EASI is a composite index with scores ranging from 0 to 72. Four AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) assessed for severity on a scale of "0" (absent) through "3" (severe). In addition, the area of AD involvement is assessed as a percentage by body area of head, trunk (including the genital area), upper extremities, and lower extremities (including the buttocks), and converted to a score of 0 to 6. In each body region, the area is expressed as 0, 1 (1% to 9%), 2 (10% to 29%), 3 (30% to 49%), 4 (50% to 69%), 5 (70% to 89%), or 6 (90% to 100%).
Time Frame: Baseline and Week 16
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dupilumab (Period 1) | Upadacitinib (Period 1)
Number analyzed (Participants) | 462 | 458
percentage of participants | 22.5 [18.7 to 26.3] | 40.8 [36.3 to 45.3]
Statistical Analysis 1: Comparison: Dupilumab (Period 1) vs Upadacitinib (Period 1); Upadacitinib (Period 1) vs Dupilumab (Period 1); Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel; Adjusted Response Rate Difference = 18.4, 95% CI 2-sided [12.5 to 24.2] — Response rate difference = Upadacitinib (Period 1) - Dupilumab (Period 1)

3. Secondary Outcome: Percentage of Participants Achieving a Worst Pruritus Numerical Rating Scale of 0 or 1 (WP-NRS 0/1) at Week 16 Among Participants With Baseline WP-NRS > 1
Description: The Worst Pruritus NRS is an assessment tool that participants used to report the intensity of their pruritus during a 24-hour recall period using an electronic hand-held device. Participants rated itch (pruritus) intensity at its worst during the past 24 hours on an 11-point scale from 0 (no itch) to 10 (worst imaginable itch).
Time Frame: Baseline and Week 16
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dupilumab (Period 1) | Upadacitinib (Period 1)
Number analyzed (Participants) | 459 | 454
percentage of participants | 15.5 [12.2 to 18.8] | 30.2 [26.0 to 34.4]
Statistical Analysis 1: Comparison: Dupilumab (Period 1) vs Upadacitinib (Period 1); Upadacitinib (Period 1) vs Dupilumab (Period 1); Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel; Adjusted Response Rate Difference = 14.7, 95% CI 2-sided [9.4 to 20.0] — Response rate difference = Upadacitinib (Period 1) - Dupilumab (Period 1)

4. Secondary Outcome: Percentage of Participants Achieving an Improvement (Reduction) in Worst Pruritus Numerical Rating Scale (WP-NRS) ≥ 4 at Week 16 Among Those With Baseline WP-NRS ≥ 4
Description: as for outcome 3
Time Frame: Baseline and Week 16
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dupilumab (Period 1) | Upadacitinib (Period 1)
Number analyzed (Participants) | 457 | 448
percentage of participants | 38.1 [33.6 to 42.5] | 54.7 [50.1 to 59.3]
Statistical Analysis 1: Comparison: Dupilumab (Period 1) vs Upadacitinib (Period 1); Upadacitinib (Period 1) vs Dupilumab (Period 1); Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel; Adjusted Response Rate Difference = 16.6, 95% CI 2-sided [10.2 to 23.0] — Response rate difference = Upadacitinib (Period 1) - Dupilumab (Period 1)

5. Secondary Outcome: Percentage of Participants Achieving a Worst Pruritus Numerical Rating Scale of 0 or 1 (WP-NRS 0/1) at Week 4 Among Participants With Baseline WP-NRS > 1
Description: as for outcome 3
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dupilumab (Period 1) | Upadacitinib (Period 1)
Number analyzed (Participants) | 459 | 454
percentage of participants | 2.8 [1.3 to 4.3] | 16.1 [12.7 to 19.5]
Statistical Analysis 1: Comparison: Dupilumab (Period 1) vs Upadacitinib (Period 1); Upadacitinib (Period 1) vs Dupilumab (Period 1); Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel; Adjusted Response Rate Difference = 13.2, 95% CI 2-sided [9.6 to 16.9] — Response rate difference = Upadacitinib (Period 1) - Dupilumab (Period 1)

6. Secondary Outcome: Percentage of Participants Achieving a Worst Pruritus Numerical Rating Scale of 0 or 1 (WP-NRS 0/1) at Week 2 Among Participants With Baseline WP-NRS > 1
Description: as for outcome 3
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dupilumab (Period 1) | Upadacitinib (Period 1)
Number analyzed (Participants) | 459 | 454
percentage of participants | 1.3 [0.3 to 2.3] | 7.7 [5.3 to 10.2]
Statistical Analysis 1: Comparison: Dupilumab (Period 1) vs Upadacitinib (Period 1); Upadacitinib (Period 1) vs Dupilumab (Period 1); Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel; Adjusted Response Rate Difference = 6.4, 95% CI 2-sided [3.8 to 9.1] — Response rate difference = Upadacitinib (Period 1) - Dupilumab (Period 1)

7. Secondary Outcome: Percentage of Participants Achieving a ≥ 90% Reduction From Baseline in Eczema Area and Severity Index Score (EASI 90) at Week 4
Description: as for outcome 2
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dupilumab (Period 1) | Upadacitinib (Period 1)
Number analyzed (Participants) | 462 | 458
percentage of participants | 9.7 [7.0 to 12.4] | 23.8 [19.9 to 27.7]
Statistical Analysis 1: Comparison: Dupilumab (Period 1) vs Upadacitinib (Period 1); Upadacitinib (Period 1) vs Dupilumab (Period 1); Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel; Adjusted Response Rate Difference = 14.1, 95% CI 2-sided [9.4 to 18.8] — Response rate difference = Upadacitinib (Period 1) - Dupilumab (Period 1)

8. Secondary Outcome: Percentage of Participants Achieving a ≥ 75% Reduction From Baseline in Eczema Area and Severity Index Score (EASI 75) at Week 2
Description: as for outcome 2
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dupilumab (Period 1) | Upadacitinib (Period 1)
Number analyzed (Participants) | 462 | 458
percentage of participants | 8.2 [5.7 to 10.7] | 26.7 [22.7 to 30.8]
Statistical Analysis 1: Comparison: Dupilumab (Period 1) vs Upadacitinib (Period 1); Upadacitinib (Period 1) vs Dupilumab (Period 1); Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel; Adjusted Response Rate Difference = 18.6, 95% CI 2-sided [13.9 to 23.3] — Response rate difference = Upadacitinib (Period 1) - Dupilumab (Period 1)

9. Secondary Outcome: Percentage of Participants Achieving a 100% Reduction From Baseline in Eczema Area and Severity Index Score (EASI 100) at Week 16
Description: as for outcome 2
Time Frame: Baseline and Week 16
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dupilumab (Period 1) | Upadacitinib (Period 1)
Number analyzed (Participants) | 462 | 458
percentage of participants | 5.6 [3.5 to 7.7] | 14.8 [11.6 to 18.1]
Statistical Analysis 1: Comparison: Dupilumab (Period 1) vs Upadacitinib (Period 1); Upadacitinib (Period 1) vs Dupilumab (Period 1); Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel; Adjusted Response Rate Difference = 9.3, 95% CI 2-sided [5.4 to 13.1] — Response rate difference = Upadacitinib (Period 1) - Dupilumab (Period 1)

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse events were collected from the time informed consent was signed through the end of the study. Median time on follow-up was for 113 days for the Dupilumab (Period 1) group; 114 days for the Upadacitinib (Period 1) group; 225 days for the Dupilumab -> Upadacitinib (Period 2) group; and 224 days for the Upadacitinib -> Upadacitinib 30 mg (Period 2) group.
Arm/Group | Dupilumab (Period 1) | Upadacitinib (Period 1) | Dupilumab -> Upadacitinib (Period 2) | Upadacitinib -> Upadacitinib 30 mg (Period 2)
All-Cause Mortality (participants affected / at risk) | 0/462 | 0/458 | 0/208 | 0/147
Serious Adverse Events (participants affected / at risk) | 5/462 | 4/458 | 0/208 | 4/147
Other Adverse Events (participants affected / at risk) | 87/462 | 156/458 | 57/208 | 30/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dupilumab (Period 1) (N=462) | Upadacitinib (Period 1) (N=458) | Dupilumab -> Upadacitinib (Period 2) (N=208) | Upadacitinib -> Upadacitinib 30 mg (Period 2) (N=147)
DRUG-INDUCED LIVER INJURY (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ANAPHYLACTIC REACTION (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
JUVENILE IDIOPATHIC ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
EPILEPSY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MIGRAINE WITHOUT AURA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DEPRESSION (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MAJOR DEPRESSION (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SUICIDAL IDEATION (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DERMATITIS ATOPIC (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
PERIPHERAL ARTERY OCCLUSION (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dupilumab (Period 1) (N=462) | Upadacitinib (Period 1) (N=458) | Dupilumab -> Upadacitinib (Period 2) (N=208) | Upadacitinib -> Upadacitinib 30 mg (Period 2) (N=147)
NASOPHARYNGITIS (Infections and infestations) | 35 (43) | 58 (74) | 18 (20) | 12 (13)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 22 (28) | 27 (33) | 12 (12) | 7 (9)
HEADACHE (Nervous system disorders) | 16 (20) | 27 (32) | 5 (5) | 1 (1)
ACNE (Skin and subcutaneous tissue disorders) | 7 (7) | 55 (56) | 14 (14) | 5 (5)
DERMATITIS ATOPIC (Skin and subcutaneous tissue disorders) | 15 (17) | 23 (24) | 12 (12) | 9 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2023-05-02): https://cdn.clinicaltrials.gov/large-docs/82/NCT05601882/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-11): https://cdn.clinicaltrials.gov/large-docs/82/NCT05601882/SAP_001.pdf